CLINICAL TRIAL: NCT00119964
Title: Weight Management for a Defined Employee Population Using an Interactive eHealth Portal
Brief Title: The Healthy Lifestyle Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 51756
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: internet based weight management tools

SUMMARY:
The purpose of this study is to determine if an internet-based intervention will be effective in improving the lifestyle and weight of an obese employee population.

The intervention will last 12 months, and includes a weight tracker, a food intake tracker, an activity tracker, a calorie balance tool, an electronic discussion board, and electronic greeting cards.

DETAILED DESCRIPTION:
The study will compare two groups over time, one of which will utilize the electronic tools, and one of which will not. The samples will be drawn from the employees of a metro-Milwaukee hospital, and will consist of obese (Body Mass Index, or BMI, of 30 or greater) employees only.

The primary outcome will be change in weight over the study time period as measured by the BMI. Secondary outcome measures will include quality of life, blood pressure, tests of blood sugar, cholesterol, presence of depression, lifestyle wellness score, health care costs and productivity.

ELIGIBILITY:
Inclusion Criteria:

* Obesity as defined by a BMI of 30 or greater
* The ability to speak and understand english
* Health insurance coverage through First Health (Aurora's employee insurance plan)
* Not currently on another formal weight management program
* Not currently taking any weight loss medications
* Not currently disabled in such a way that participation would be precluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2004-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
change in body mass index

SECONDARY OUTCOMES:
quality of life
blood pressure
hemoglobin A1c
total cholesterol
HDL cholesterol
HANDS depression score
wellness score on Summex Health Risk Appraisal
health care costs
unscheduled paid time off

CONTACTS AND LOCATIONS:
Overall Officials: Alison Lux, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Milwaukee, Wisconsin, United States